CLINICAL TRIAL: NCT03277664
Title: The Effect of Electronic Monitoring Combined With Weekly Feedback and Reminders on Adherence to Inhaled Corticosteroids in Infants and Younger Children With Asthma: a Randomized Controlled Trial
Brief Title: Electronic Monitoring Combined With Weekly Feedback and Reminders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: ESR-15-11001
Record Dates: First submitted 2017-09-06; First posted 2017-09-11 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Asthma
Keywords: pediatric; asthma adherence; electronic device
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: The Study of Asthma Adherence study was a multicentre, single-blind, parallel group randomised controlled trial, with an allocation ratio of 1:1.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, the caregivers of the participants and follow-up nurse were not blinded. But the doctors and statisticians were blinded. Both in the intervention group and control group, adherence data were not available to clinicians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): All the device-monitored adherence data from the previous week were downloaded from the background database and calculated by a qualified asthma nurse. Through free IMS (WeChat; Tencent, Shenzhen, CHN) available on mobile, the nurse offered feedback to the caregivers weekly according to the adherence rate and reminded them to keep taking the ICS. Caregivers were asked monthly "Has our child inhaled the medicine according to the doctor's instructions?" and "How about the frequency?" by telephone.
  Interventions: Behavioral: intervention group
- control group (No Intervention): All the device-monitored adherence data were downloaded from the background database and calculated weekly. However, feedback and reminders were not given to the caregivers. Caregivers were also asked monthly "Has our child inhaled the medicine according to the doctor's instructions?" and "How about the frequency?" by telephone.

INTERVENTIONS:
Behavioral: intervention group — All the device-monitored adherence data from the previous week were downloaded from the background database and calculated by a qualified asthma nurse. Through free IMS (WeChat; Tencent, Shenzhen, CHN) available on mobile, the nurse offered feedback to the caregivers weekly according to the adherence rate and reminded them to keep taking the ICS. Caregivers were asked monthly "Has our child inhaled the medicine according to the doctor's instructions?" and "How about the frequency?" by telephone.
  Arms: intervention group

SUMMARY:
A total of 96 recruited children (aged 6 months to 3 years) with mild or moderate persistent asthma who were on regular inhaled corticosteroids (ICS) were randomly allocated to receive electronic monitoring combined with instant messaging software -based weekly feeding back adherence and reminders to keep taking the ICS (intervention group) and to receive electronic monitoring only (control group). The device-monitored adherence rates and caregiver-reported adherence rates were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. patients having mild or moderate persistent asthma
2. 6 months-3 years
3. taking regular inhaled steroids, with no change in their medication in the last month.

Exclusion Criteria:

Participants who had severe persistent asthma or another respiratory disease or did not live in Shanghai were excluded.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
device monitored adherence rate | up to 6 months
  The primary outcome of the study was change in the adherence rate monitored by the electronic device for 6 consecutive months. This adherence rate was calculated as the number of device recorded times /number of total times prescribed × 100%.

SECONDARY OUTCOMES:
caregiver-reported adherence rate | up to 6 months
  The secondary outcomes for the study were the caregiver-reported adherence rate and the difference between device-monitored and caregiver-reported adherence rates for 6 consecutive months. The caregiver-reported adherence rate was recorded on a monthly basis. It was offered by the caregivers of patients through answering the questions "Has our child inhaled the medicine according to the doctor's instructions" and "How about the frequency". The device-monitored and caregiver-reported adherence rates were compared monthly.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai children's medical center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen J, Xu J, Zhao L, Zhang J, Yin Y, Zhang F. The effect of electronic monitoring combined with weekly feedback and reminders on adherence to inhaled corticosteroids in infants and younger children with asthma: a randomized controlled trial. Allergy Asthma Clin Immunol. 2020 Jul 29;16:68. doi: 10.1186/s13223-020-00466-6. eCollection 2020. PMID 32922454